CLINICAL TRIAL: NCT07354425
Title: Pneumococcal Community-Acquired Pneumonia Requiring Hospitalization Among Colombian Adults (Pneumo-CAP Colombia)
Brief Title: Pneumococcal Community-Acquired Pneumonia Requiring Hospitalization Among Colombian Adults
Acronym: PneumoCAP
Status: Completed | Type: Observational
Sponsor: Universidad de la Sabana (Other)
Collaborators: Clínica Universidad de La Sabana (Unknown); Universidad de La Sabana, Colombia (Unknown)
Responsible Party: Principal Investigator, Luis Felipe Reyes, MD, PhD, MSc Principal Investigator, Universidad de la Sabana
Other Study IDs: MED-357-2023
Record Dates: First submitted 2025-11-27; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Community Acquired Pneumonia (CAP); Pneumococcal Pneumonia
Keywords: Pneumo-CAP; Community Acquired Pneumonia; CAP; Pneumococcal Pneumonia; Colombia
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumonia, Pneumococcal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Biospecimen Retention: Samples With DNA — Blood Urine Sputum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pneumococcal Community-Acquired Pneumonia Requiring Hospitalization Among Adults in Colombia (Pneumo-CAP Colombia)

This study aims to learn more about pneumococcal community-acquired pneumonia (CAP) caused by Streptococcus pneumoniae among adults hospitalized in 11 hospitals in the Sabana Centro region of Colombia. The study will describe the characteristics of adults with CAP, estimate pneumococcal CAP prevalence in the area, and examine the specific serotypes of S. pneumoniae causing this infection. This research is essential for understanding which microorganism is the most prevalent cause of CAP in the region, whether pneumococcal vaccines included in governmental vaccination programs protect adults, which specific pneumococcal serotypes are circulating, and which available vaccine will best protect people against pneumococcal CAP.

The study will be conducted at 11 hospitals in the Sabana Centro region and will collect data over 2 years. The study will gather detailed information on each patient's condition, including symptoms, medical history, and outcomes such as death or the need for intensive care.

DETAILED DESCRIPTION:
This prospective, multicenter surveillance study aims to provide a detailed understanding of pneumococcal community-acquired pneumonia (CAP), a leading cause of hospitalization and mortality, in adults in the Sabana Centro region of Colombia. Pneumococcal CAP, caused by the bacterium Streptococcus pneumoniae, remains a significant global health burden despite widespread vaccination programs. The study will investigate the incidence, prevalence, and serotype distribution of pneumococcal CAP, with a particular focus on strains included in the 15-valent pneumococcal conjugate vaccine (PCV15).

The study's objectives will help inform future vaccine development, public health policies, and the clinical management of pneumococcal infections in adult populations, particularly in low- and middle-income countries (LMICs), where vaccine coverage and disease burden remain concerns.

Study Goals and Objectives:

The study has four primary objectives:

1. To describe the demographic and clinical characteristics of adults ≥18 years hospitalized with pneumococcal CAP in the Sabana Centro region, including both bacteremic and non-bacteremic cases of the infection.
2. To determine the prevalence of pneumococcal CAP among patients requiring hospitalization for CAP in the Sabana Centro region of Colombia.
3. To determine the prevalence of pneumococcal serotypes included in the PCV15 vaccine in hospitalized adults with pneumococcal CAP, including both bacteremic and non-bacteremic cases.
4. To estimate the incidence of pneumococcal CAP that requires hospitalization and the contribution of PCV15 serotypes to the disease burden in the region.

   The study will also explore secondary objectives, including the association between pneumococcal positivity and severe clinical outcomes like ICU admission, mechanical ventilation, vasopressor use, and mortality.

   Study Design:

   This is a prospective, observational, multicenter study with active surveillance. The research will take place at 11 hospitals across the Sabana Centro region, including both public and private institutions. The study will collect data over two years, with a recruitment period of one year and a follow-up period of up to three months post-discharge.

   Inclusion and Exclusion Criteria:

   Inclusion Criteria:

   -1. Age ≥ 18 years old.

   -2. Hospitalized at one of the hospitals of Sabana Centro Region, including both in-patient and observation status stay.

   -3.Clinical signs and/or symptoms of an acute respiratory illness, as defined by ≥ 1 of the following:

   -New or worsening shortness of breath in the past 7 days

   -New or worsening cough in the past 7 days

   -New or worsening sputum production in the past 7 days

   -New or worsening chest pain in the past 7 days

   -Tachypnea to respiratory rate ≥ 22 breaths/min, not known to be chronic

   -Hypoxia to SpO2 ≤ 92% not known to be chronic

   -Initiation of invasive or non-invasive mechanical ventilation.

   -4. Clinical signs and/or symptoms of an acute infection, as defined by ≥ 1 of the following:

   -Body temperature ≥ 38º C (100.4º F) or ≤ 35.5º C (95.9º F)

   -Reported fever, chills, or feeling feverish at home without explicit documentation of a fever within the past 7 days

   -White blood cell count > 10.7 or < 3.9 thousand cells/mcL-C-reactive protein > 10 mg/L
   * Altered mental status
   * 5. Radiologic evidence of pneumonia interpreted by a radiologist, defined as ≥ 1 of the following findings on chest x-ray (CXR), computed tomography (CT), or lung ultrasound completed within 48 hours before or after hospital admission:
   * Pulmonary infiltrate not known to be chronic
   * Pulmonary opacity is not known to be chronic (including ground-glass opacities on CT)
   * Pulmonary consolidation is not known to be

   Exclusion Criteria:

   -1. Enrollment in this study within the past 90 days.

   -2. Development of pneumonia (as defined in the inclusion criteria) more than 48 hours after hospital admission (pneumonia developed 48 hours after admission will be considered hospital-acquired pneumonia).

   -3. Inability to obtain consent from patient or surrogate for this study within 48 hours of hospital admission (including time at a transferring hospital before admission at a study hospital).

   -4. Inability or unwillingness of the patient to provide any of the samples (Blood, Urine, and Sputum) within 48 hours of hospital admission (including time at a transferring hospital before admission at a study hospital).

   -5. Non-pneumonia illness completely explains the patient's acute symptoms. Alternative non-pneumonia illnesses could include pulmonary embolism, acute heart failure, lung cancer, and pulmonary hemorrhage.

   o- Key Outcomes and Data Collection:

   The study will track multiple outcomes, including:

   o- Incidence of pneumococcal CAP (overall, and by specific serotypes included in PCV15).

   o- Prevalence of pneumococcal serotypes, particularly those contained in PCV15.

   o- Clinical outcomes such as:

   o Mortality (hospital mortality and 3-month post-discharge mortality)

   o ICU admission

   o Need for invasive mechanical ventilation

   o Use of vasopressors

   o Duration of hospital and ICU stay

   o- Quality of life measures using the EQ-5D-5L and mMRC scales, assessed at baseline, 1 month, and 3 months post-discharge.

   o- Laboratory Tests and Procedures:

   The study will use a combination of diagnostic methods to detect S. pneumoniae and characterize the pneumococcal strains involved, including:

   o Urine antigen tests.

   o Blood cultures.
   * Sputum cultures.
   * Real-time PCR for molecular detection of S. pneumoniae in blood and sputum samples.

   In addition, the study will collect data on the antimicrobial resistance patterns of the isolated pneumococcal strains, evaluating resistance to penicillins, macrolides, and other antibiotic classes.

   o-Data Management and Analysis: All data will be collected electronically through the RedCap platform, a secure, web-based system. The data will be analyzed using descriptive statistics for demographic and clinical characteristics, as well as incidence and prevalence rates of pneumococcal CAP. Multivariate regression models will be used to assess associations between pneumococcal infection and clinical outcomes, while adjusting for potential confounders such as age, sex, comorbidities, and vaccination status.

   o- Follow-Up: Patients will be followed up by phone at 1 and 3 months post-discharge to evaluate long-term outcomes, including survival, functional recovery, and quality of life. This follow-up is crucial for understanding the long-term burden of pneumococcal CAP and the potential impact of vaccination.

   o- Study Timeline and Sample Size: The study is expected to run for 2 years. The study will include all eligible patients hospitalized during this time, and the number of qualifying cases observed will determine the sample size.

   o- Ethical Considerations and Confidentiality: The study will be conducted in accordance with ethical guidelines for human research and will obtain approval from institutional review boards (IRBs) at all participating hospitals. Informed consent will be obtained from all patients (or their legal representatives) before enrollment. All patient data will be kept confidential, and participants will be identified only by a study-specific ID.

   o- Study Significance and Expected Impact: This study is the first of its kind in Colombia to comprehensively evaluate the incidence, prevalence, and clinical outcomes of pneumococcal CAP in adults. The findings will provide crucial data on the pneumococcal serotypes circulating in the region, informing vaccine policy and the potential introduction of new pneumococcal vaccines, such as PCV15, into the Colombian adult population. The study also aims to address the significant knowledge gap in the epidemiology of pneumococcal infections in LMICs, where data on adult pneumococcal CAP is limited.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age ≥ 18 years old.
* (2) Hospitalized at one of the hospitals of Sabana Centro Region, including both in-patient and observation status stay.
* (3) Clinical signs and/or symptoms of an acute respiratory illness, as defined by ≥ 1 of the
* following:
* -New or worsening shortness of breath in the past 7 days
* -New or worsening cough in the past 7 days
* -New or worsening sputum production in the past 7 days
* -New or worsening chest pain in the past 7 days
* -Tachypnea to respiratory rate ≥ 22 breaths/min, not known to be chronic
* -Hypoxia to SpO2 ≤ 92% not known to be chronic
* -Initiation of invasive or non-invasive mechanical ventilation
* (4) Clinical signs and/or symptoms of an acute infection, as defined by ≥ 1 of the following:
* -Body temperature ≥ 38º C (100.4º F) or ≤ 35.5º C (95.9º F)
* -Reported fever, chills, or feeling feverish at home without explicit documentation of a fever within the past 7 days
* -White blood cell count > 10.7 or < 3.9 thousand cells/mcL-C-reactive protein > 10 mg/L
* -Altered mental status
* (5) Radiologic evidence of pneumonia interpreted by a radiologist, defined as ≥ 1 of the following findings on chest x-ray (CXR), computed tomography (CT), or lung ultrasound completed within 48 hours before or after hospital admission:
* -Pulmonary infiltrate not known to be chronic
* -Pulmonary opacity is not known to be chronic (including ground-glass opacities on CT)
* -Pulmonary consolidation is not known to be

Exclusion Criteria:

* (1) Enrollment in this study within the past 90 days.
* (2) Development of pneumonia (as defined in the inclusion criteria) more than 48 hours after hospital admission (pneumonia developed 48 hours after admission will be considered hospital-acquired pneumonia).
* (3) Inability to obtain consent from patient or surrogate for this study within 48 hours of hospital admission (including time at a transferring hospital before admission at a study hospital).
* (4) Inability or unwillingness of the patient to provide any of the samples (Blood, Urine, and Sputum) within 48 hours of hospital admission (including time at a transferring hospital before admission at a study hospital).
* (5) Non-pneumonia illness completely explains the patient's acute symptoms. Alternative non-pneumonia illnesses could include pulmonary embolism, acute heart failure, lung cancer, and pulmonary hemorrhage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adults aged 18 years or older hospitalized with community-acquired pneumonia (CAP) in the Sabana Centro region of Colombia. This region includes 11 municipalities around Bogotá and represents a diverse socio-economic and demographic population with a well-organized healthcare system.
Sampling Method: Non-Probability Sample
Enrollment: 688 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
Incidence of Pneumococcal Community-Acquired Pneumonia (CAP) | The incidence will be measured throughout the whole study period (from study start to study end), with cases recorded at the time of hospital admission for CAP. (2 years)(Jun-2022 to Nov-2025)
  This outcome captures how many adults are hospitalized with community-acquired pneumonia caused by Streptococcus pneumoniae, including both bacteremic (positive blood culture) and non-bacteremic cases (positive respiratory sample, urinary antigen test, or PCR).
  How it will be measured
  Pneumococcal CAP cases will be identified through routinely collected microbiological results:
  Blood cultures Respiratory cultures (sputum, BAL, tracheal aspirate) Urinary pneumococcal antigen test PCR/NAAT panels detecting S. pneumoniae All confirmed cases will be counted and divided by the total number of CAP hospitalizations (or by the catchment population, if applicable) to calculate the incidence.
Prevalence of Pneumococcal Serotypes | Serotypes will be assessed at the time of hospitalization, and the prevalence will be evaluated across the entire study period. (2 years, Jun-2022 until Nov-2025)
  This outcome describes the frequency with which pneumococcal serotypes covered by the 15-valent conjugate vaccine (PCV15) appear among adults hospitalized with community-acquired pneumonia.
  How it will be measured All patients with pneumococcal CAP who undergo serotyping will be reviewed. Each serotype identified will be classified as either a PCV15 serotype or a non-PCV15 serotype. The prevalence will be determined by counting the number of pneumococcal CAP cases caused by serotypes included in PCV15, compared with the total number of cases with available serotype information.
Prevalence of Pneumococcal CAP Among Hospitalized Adults | Pneumococcal CAP cases will be identified at the time of hospital admission, and prevalence will be assessed for the entire study period.(2 years, Jun-2022 until Nov-2025)
  This outcome describes the prevalence of community-acquired pneumococcal pneumonia among adults requiring hospitalization.
  How it will be measured All hospitalized adults diagnosed with CAP will be reviewed to determine which cases have laboratory confirmation of Streptococcus pneumoniae through blood cultures, respiratory samples, urinary antigen testing, or molecular assays. The prevalence will be determined by counting the number of CAP cases identified as pneumococcal among all CAP hospitalizations.

SECONDARY OUTCOMES:
Severity of Pneumococcal CAP | Recorded on day 1 ( baseline) and/or at ICU admission when applicable.
  This outcome describes the clinical severity of pneumococcal community-acquired pneumonia among hospitalized adults, based on routinely used severity assessment tools.
  How it will be measured
  Severity will be determined using any of the three validated clinical scales routinely used by the treating clinician, and patients will be classified as having severe or non-severe disease according to the score applied:
  Pneumonia Severity Index (PSI) Range: Class I to Class V (0 to >130 points). Higher scores indicate worse severity and higher mortality risk. CURB-65 Score (Confusion, Urea, Respiratory rate, Blood pressure, Age ≥65) Range: 0 to 5 points. Higher scores indicate greater severity and higher mortality risk. Severe Community-Acquired Pneumonia Criteria (American Thoracic Society/Infectious Diseases Society of America) Definition: Severe CAP is identified by 1 major criterion or ≥3 minor criteria. Meeting criteria indicates higher severity and need for intensive care.
Mortality | from recruitment until 3 months post-discharge
  In-hospital mortality and 3-month post-discharge mortality
ICU Admission | Recorded on day of ICU admission (during index hospitalization)
  This outcome captures whether adults hospitalized with CAP require admission to an intensive care unit at any point during their hospitalization, reflecting higher disease severity and need for advanced organ support.
  How it will be measured ICU admission will be determined through routine hospital records, documenting whether the patient was admitted to an ICU (medical, surgical, or mixed) during the index hospitalization. This includes admissions occurring directly from the emergency department or later during the hospital stay, up to discharge.
Variation in Quality of Life | Recorded on day 1 ( baseline) and on day 27 after discharge and day 90 after discharge (From recruitment until 3 month post-discharge)
  This outcome evaluates changes in quality of life among adults hospitalized with CAP, using the standardized EQ-5D-5L instrument, which measures health status across five domains.
  How it will be measured Quality of life will be assessed using the EuroQol 5-Dimension 5-Level (EQ-5D-5L) scale, which includes five domains (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each scored from Level 1 (no problems) to Level 5 (extreme problems).
  The EQ-5D-5L also includes a visual analogue scale (EQ-VAS) ranging from 0 (worst imaginable health) to 100 (best imaginable health).
  Higher scores on the descriptive system indicate worse health, while higher VAS values indicate better perceived health.
  Variation will be assessed by comparing scores at different time points, based on when the tool is administered.
Dyspnea persistence | Dyspnea will be assessed at the time points defined on Day 1, Day 27 after discharge, and Day 90 after discharge. From baseline until 3 months post-discharge.
  This outcome evaluates whether adults hospitalized with CAP continue to experience shortness of breath after the acute illness, using a standardized measure of breathlessness severity.
  How it will be measured Dyspnea will be assessed using the modified Medical Research Council (mMRC) Dyspnea Scale, which ranges from Grade 0 to Grade 4.
  Grade 0: Breathlessness only with strenuous exercise Grade 1: Shortness of breath when hurrying or walking up a slight hill Grade 2: Walks slower than peers or must stop when walking at own pace Grade 3: Stops for breath after walking ~100 meters Grade 4: Too breathless to leave the house or breathless when dressing Higher mMRC grades indicate worse dyspnea. Persistence will be determined by comparing dyspnea scores across relevant follow-up time points.

CONTACTS AND LOCATIONS:
Overall Officials: Luis F Reyes, MD,PhD, MsC, Principal Investigator — Universidad de la Sabana; Cristian C Serrano, MD, cPhD, Principal Investigator — Clinica Universidad de La Sabana
Locations (11):
- Colombia (11):
  - Clinica de Marly Jorge Cavelier Gaviria SAS, Chía, Cundinamarca
  - Clinica Universidad de La Sabana, Chía, Cundinamarca
  - ESE Hospital San Antonio de Chia, Chía, Cundinamarca
  - Centro Medico San Luis Clinica Quirurgica SAS, Cajicá
  - ESE Hospital San Vicente de Paul Nemocon, Nemocón
  - ESE Hospital divino Salvador Sopo, Sopó
  - ESE Hospital Nuestra Señora del Carmen de Tabio, Tabio
  - ESE Hospital Santa Rosa de Tenjo, Tenjo
  - Hospital Nuestra Señora del Transito de Tocancipa, Tocancipá
  - Hospital Universitario de la Samaritana Regional, Zipaquirá
  - Hospital Universitario de la Samaritana sede Funcional, Zipaquirá

IPD SHARING:
Plan to Share IPD: Undecided
The decision regarding the sharing of individual participant data has not yet been finalized. IPD availability will depend on ethical approvals, institutional policies, and data-governance requirements across participating sites.

REFERENCES:
- [Background] Kung HC, Hoyert DL, Xu J, Murphy SL. Deaths: final data for 2005. Natl Vital Stat Rep. 2008 Apr 24;56(10):1-120. PMID 18512336
- [Background] Agency for Healthcare Research and Quality. Pneumonia is the Most Common Reason for Hospitalization. http://www.ahrq.gov/research/sep08/0908RA40.htm Accessed: 31 May 2011.
- [Background] Self WH, Grijalva CG, Zhu Y, McNaughton CD, Barrett TW, Collins SP, Storrow AB, Griffin MR. Rates of emergency department visits due to pneumonia in the United States, July 2006-June 2009. Acad Emerg Med. 2013 Sep;20(9):957-60. doi: 10.1111/acem.12203. Epub 2013 Aug 27. PMID 24033659
- [Background] Grijalva CG, Nuorti JP, Arbogast PG, Martin SW, Edwards KM, Griffin MR. Decline in pneumonia admissions after routine childhood immunisation with pneumococcal conjugate vaccine in the USA: a time-series analysis. Lancet. 2007 Apr 7;369(9568):1179-86. doi: 10.1016/S0140-6736(07)60564-9. PMID 17416262
- [Background] Leal AL, Camacho G, Montañez A, Varon F, Alvarez C, Valderrama S, et al. 1628. Clinical, Epidemiological and Microbiological Characterization of Invasive Streptococcus pneumoniae Disease in Hospitalized Adults from 5 Tertiary Hospitals in Bogotá, Colombia: A Descriptive Study, Open Forum Infectious Diseases, Volume 6, Issue Supplement_2, October 2019, Pages S593-S594.
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Severiche-Bueno DF, Severiche-Bueno DF, Bastidas A, Caceres EL, Silva E, Lozada J, Gomez S, Vargas H, Viasus D, Reyes LF. Burden of invasive pneumococcal disease (IPD) over a 10-year period in Bogota, Colombia. Int J Infect Dis. 2021 Apr;105:32-39. doi: 10.1016/j.ijid.2021.02.031. Epub 2021 Feb 11. PMID 33582374
- [Background] Jain S, Williams DJ, Arnold SR, Ampofo K, Bramley AM, Reed C, Stockmann C, Anderson EJ, Grijalva CG, Self WH, Zhu Y, Patel A, Hymas W, Chappell JD, Kaufman RA, Kan JH, Dansie D, Lenny N, Hillyard DR, Haynes LM, Levine M, Lindstrom S, Winchell JM, Katz JM, Erdman D, Schneider E, Hicks LA, Wunderink RG, Edwards KM, Pavia AT, McCullers JA, Finelli L; CDC EPIC Study Team. Community-acquired pneumonia requiring hospitalization among U.S. children. N Engl J Med. 2015 Feb 26;372(9):835-45. doi: 10.1056/NEJMoa1405870. PMID 25714161
- [Background] Moore MR, Link-Gelles R, Schaffner W, Lynfield R, Lexau C, Bennett NM, Petit S, Zansky SM, Harrison LH, Reingold A, Miller L, Scherzinger K, Thomas A, Farley MM, Zell ER, Taylor TH Jr, Pondo T, Rodgers L, McGee L, Beall B, Jorgensen JH, Whitney CG. Effect of use of 13-valent pneumococcal conjugate vaccine in children on invasive pneumococcal disease in children and adults in the USA: analysis of multisite, population-based surveillance. Lancet Infect Dis. 2015 Mar;15(3):301-9. doi: 10.1016/S1473-3099(14)71081-3. Epub 2015 Feb 3. PMID 25656600
- [Background] Griffin MR, Zhu Y, Moore MR, Whitney CG, Grijalva CG. U.S. hospitalizations for pneumonia after a decade of pneumococcal vaccination. N Engl J Med. 2013 Jul 11;369(2):155-63. doi: 10.1056/NEJMoa1209165. PMID 23841730
- [Background] Jain S, Self WH, Wunderink RG, Fakhran S, Balk R, Bramley AM, Reed C, Grijalva CG, Anderson EJ, Courtney DM, Chappell JD, Qi C, Hart EM, Carroll F, Trabue C, Donnelly HK, Williams DJ, Zhu Y, Arnold SR, Ampofo K, Waterer GW, Levine M, Lindstrom S, Winchell JM, Katz JM, Erdman D, Schneider E, Hicks LA, McCullers JA, Pavia AT, Edwards KM, Finelli L; CDC EPIC Study Team. Community-Acquired Pneumonia Requiring Hospitalization among U.S. Adults. N Engl J Med. 2015 Jul 30;373(5):415-27. doi: 10.1056/NEJMoa1500245. Epub 2015 Jul 14. PMID 26172429
- [Background] Said MA, Johnson HL, Nonyane BA, Deloria-Knoll M, O'Brien KL; AGEDD Adult Pneumococcal Burden Study Team; Andreo F, Beovic B, Blanco S, Boersma WG, Boulware DR, Butler JC, Carratala J, Chang FY, Charles PG, Diaz AA, Dominguez J, Ehara N, Endeman H, Falco V, Falguera M, Fukushima K, Garcia-Vidal C, Genne D, Guchev IA, Gutierrez F, Hernes SS, Hoepelman AI, Hohenthal U, Johansson N, Kolek V, Kozlov RS, Lauderdale TL, Marekovic I, Masia M, Matta MA, Miro O, Murdoch DR, Nuermberger E, Paolini R, Perello R, Snijders D, Plecko V, Sorde R, Stralin K, van der Eerden MM, Vila-Corcoles A, Watt JP. Estimating the burden of pneumococcal pneumonia among adults: a systematic review and meta-analysis of diagnostic techniques. PLoS One. 2013;8(4):e60273. doi: 10.1371/journal.pone.0060273. Epub 2013 Apr 2. PMID 23565216
- [Background] Wunderink RG, Self WH, Anderson EJ, Balk R, Fakhran S, Courtney DM, Qi C, Williams DJ, Zhu Y, Whitney CG, Moore MR, Bramley A, Jain S, Edwards KM, Grijalva CG. Pneumococcal Community-Acquired Pneumonia Detected by Serotype-Specific Urinary Antigen Detection Assays. Clin Infect Dis. 2018 May 2;66(10):1504-1510. doi: 10.1093/cid/cix1066. PMID 29342250
- [Background] LeBlanc JJ, ElSherif M, Ye L, MacKinnon-Cameron D, Li L, Ambrose A, Hatchette TF, Lang AL, Gillis H, Martin I, Andrew MK, Boivin G, Bowie W, Green K, Johnstone J, Loeb M, McCarthy A, McGeer A, Moraca S, Semret M, Stiver G, Trottier S, Valiquette L, Webster D, McNeil SA; Serious Outcomes Surveillance (SOS) Network of the Canadian Immunization Research Network (CIRN). Burden of vaccine-preventable pneumococcal disease in hospitalized adults: A Canadian Immunization Research Network (CIRN) Serious Outcomes Surveillance (SOS) network study. Vaccine. 2017 Jun 22;35(29):3647-3654. doi: 10.1016/j.vaccine.2017.05.049. Epub 2017 May 26. PMID 28554501
- [Background] Pilishvili T, Lexau C, Farley MM, Hadler J, Harrison LH, Bennett NM, Reingold A, Thomas A, Schaffner W, Craig AS, Smith PJ, Beall BW, Whitney CG, Moore MR; Active Bacterial Core Surveillance/Emerging Infections Program Network. Sustained reductions in invasive pneumococcal disease in the era of conjugate vaccine. J Infect Dis. 2010 Jan 1;201(1):32-41. doi: 10.1086/648593. PMID 19947881
- [Background] Demczuk WH, Martin I, Griffith A, Lefebvre B, McGeer A, Lovgren M, Tyrrell GJ, Desai S, Sherrard L, Adam H, Gilmour M, Zhanel GG; Toronto Bacterial Diseases Network; Canadian Public Health Laboratory Network. Serotype distribution of invasive Streptococcus pneumoniae in Canada after the introduction of the 13-valent pneumococcal conjugate vaccine, 2010-2012. Can J Microbiol. 2013 Dec;59(12):778-88. doi: 10.1139/cjm-2013-0614. Epub 2013 Oct 21. PMID 24313450
- [Background] Waight PA, Andrews NJ, Ladhani SN, Sheppard CL, Slack MP, Miller E. Effect of the 13-valent pneumococcal conjugate vaccine on invasive pneumococcal disease in England and Wales 4 years after its introduction: an observational cohort study. Lancet Infect Dis. 2015 May;15(5):535-43. doi: 10.1016/S1473-3099(15)70044-7. Epub 2015 Mar 20. PMID 25801458
- [Background] van der Linden M, Falkenhorst G, Perniciaro S, Imohl M. Effects of Infant Pneumococcal Conjugate Vaccination on Serotype Distribution in Invasive Pneumococcal Disease among Children and Adults in Germany. PLoS One. 2015 Jul 1;10(7):e0131494. doi: 10.1371/journal.pone.0131494. eCollection 2015. PMID 26132078
- [Background] American Thoracic Society; Infectious Diseases Society of America. Guidelines for the management of adults with hospital-acquired, ventilator-associated, and healthcare-associated pneumonia. Am J Respir Crit Care Med. 2005 Feb 15;171(4):388-416. doi: 10.1164/rccm.200405-644ST. No abstract available. PMID 15699079
- [Background] Self WH, Wunderink RG, Williams DJ, Barrett TW, Baughman AH, Grijalva CG. Comparison of clinical prediction models for resistant bacteria in community-onset pneumonia. Acad Emerg Med. 2015 Jun;22(6):730-40. doi: 10.1111/acem.12672. Epub 2015 May 20. PMID 25996620
- [Background] Kalil AC, Metersky ML, Klompas M, Muscedere J, Sweeney DA, Palmer LB, Napolitano LM, O'Grady NP, Bartlett JG, Carratala J, El Solh AA, Ewig S, Fey PD, File TM Jr, Restrepo MI, Roberts JA, Waterer GW, Cruse P, Knight SL, Brozek JL. Management of Adults With Hospital-acquired and Ventilator-associated Pneumonia: 2016 Clinical Practice Guidelines by the Infectious Diseases Society of America and the American Thoracic Society. Clin Infect Dis. 2016 Sep 1;63(5):e61-e111. doi: 10.1093/cid/ciw353. Epub 2016 Jul 14. PMID 27418577
- [Background] Grijalva CG, Wunderink RG, Zhu Y, Williams DJ, Balk R, Fakhran S, Courtney DM, Anderson EJ, Qi C, Trabue C, Pavia AT, Moore MR, Jain S, Edwards KM, Self WH. In-Hospital Pneumococcal Polysaccharide Vaccination Is Associated With Detection of Pneumococcal Vaccine Serotypes in Adults Hospitalized for Community-Acquired Pneumonia. Open Forum Infect Dis. 2015 Sep 19;2(4):ofv135. doi: 10.1093/ofid/ofv135. eCollection 2015 Dec. PMID 26512357
- [Background] Upchurch CP, Grijalva CG, Wunderink RG, Williams DJ, Waterer GW, Anderson EJ, Zhu Y, Hart EM, Carroll F, Bramley AM, Jain S, Edwards KM, Self WH. Community-Acquired Pneumonia Visualized on CT Scans but Not Chest Radiographs: Pathogens, Severity, and Clinical Outcomes. Chest. 2018 Mar;153(3):601-610. doi: 10.1016/j.chest.2017.07.035. Epub 2017 Aug 9. PMID 28802696
- [Background] Fine MJ, Auble TE, Yealy DM, Hanusa BH, Weissfeld LA, Singer DE, Coley CM, Marrie TJ, Kapoor WN. A prediction rule to identify low-risk patients with community-acquired pneumonia. N Engl J Med. 1997 Jan 23;336(4):243-50. doi: 10.1056/NEJM199701233360402. PMID 8995086
- [Background] Lim WS, van der Eerden MM, Laing R, Boersma WG, Karalus N, Town GI, Lewis SA, Macfarlane JT. Defining community acquired pneumonia severity on presentation to hospital: an international derivation and validation study. Thorax. 2003 May;58(5):377-82. doi: 10.1136/thorax.58.5.377. PMID 12728155
- [Background] Mandell LA, Wunderink RG, Anzueto A, Bartlett JG, Campbell GD, Dean NC, Dowell SF, File TM Jr, Musher DM, Niederman MS, Torres A, Whitney CG; Infectious Diseases Society of America; American Thoracic Society. Infectious Diseases Society of America/American Thoracic Society consensus guidelines on the management of community-acquired pneumonia in adults. Clin Infect Dis. 2007 Mar 1;44 Suppl 2(Suppl 2):S27-72. doi: 10.1086/511159. No abstract available. PMID 17278083
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Buurman BM, Hoogerduijn JG, de Haan RJ, Abu-Hanna A, Lagaay AM, Verhaar HJ, Schuurmans MJ, Levi M, de Rooij SE. Geriatric conditions in acutely hospitalized older patients: prevalence and one-year survival and functional decline. PLoS One. 2011;6(11):e26951. doi: 10.1371/journal.pone.0026951. Epub 2011 Nov 14. PMID 22110598
- [Background] Inouye SK, Rushing JT, Foreman MD, Palmer RM, Pompei P. Does delirium contribute to poor hospital outcomes? A three-site epidemiologic study. J Gen Intern Med. 1998 Apr;13(4):234-42. doi: 10.1046/j.1525-1497.1998.00073.x. PMID 9565386
- [Background] Collin C, Wade DT, Davies S, Horne V. The Barthel ADL Index: a reliability study. Int Disabil Stud. 1988;10(2):61-3. doi: 10.3109/09638288809164103. PMID 3403500
- [Background] Needham DM, Sepulveda KA, Dinglas VD, Chessare CM, Friedman LA, Bingham CO 3rd, Turnbull AE. Core Outcome Measures for Clinical Research in Acute Respiratory Failure Survivors. An International Modified Delphi Consensus Study. Am J Respir Crit Care Med. 2017 Nov 1;196(9):1122-1130. doi: 10.1164/rccm.201702-0372OC. PMID 28537429
- [Background] Colantuoni E, Scharfstein DO, Wang C, Hashem MD, Leroux A, Needham DM, Girard TD. Statistical methods to compare functional outcomes in randomized controlled trials with high mortality. BMJ. 2018 Jan 3;360:j5748. doi: 10.1136/bmj.j5748. PMID 29298779
- [Background] EuroQol. EQ-5D-5L Valuation, Crosswalk Index Value Calculator. Available at: https://euroqol.org/eq-5d- instruments/eq-5d-5l-about/valuation/crosswalk-index-valuecalculator/ Accessed 25 May 2018.
- [Background] van Hout B, Janssen MF, Feng YS, Kohlmann T, Busschbach J, Golicki D, Lloyd A, Scalone L, Kind P, Pickard AS. Interim scoring for the EQ-5D-5L: mapping the EQ-5D-5L to EQ-5D-3L value sets. Value Health. 2012 Jul-Aug;15(5):708-15. doi: 10.1016/j.jval.2012.02.008. Epub 2012 May 24. PMID 22867780
- [Background] Dowdy DW, Eid MP, Sedrakyan A, Mendez-Tellez PA, Pronovost PJ, Herridge MS, Needham DM. Quality of life in adult survivors of critical illness: a systematic review of the literature. Intensive Care Med. 2005 May;31(5):611-20. doi: 10.1007/s00134-005-2592-6. Epub 2005 Apr 1. PMID 15803303
- [Background] Dorman PJ, Slattery J, Farrell B, Dennis MS, Sandercock PA. A randomised comparison of the EuroQol and Short Form-36 after stroke. United Kingdom collaborators in the International Stroke Trial. BMJ. 1997 Aug 23;315(7106):461. doi: 10.1136/bmj.315.7106.461. No abstract available. PMID 9284664
- [Background] Angus DC, Carlet J; 2002 Brussels Roundtable Participants. Surviving intensive care: a report from the 2002 Brussels Roundtable. Intensive Care Med. 2003 Mar;29(3):368-77. doi: 10.1007/s00134-002-1624-8. Epub 2003 Jan 21. PMID 12536269
- [Background] Needham DM, Colantuoni E, Mendez-Tellez PA, Dinglas VD, Sevransky JE, Dennison Himmelfarb CR, Desai SV, Shanholtz C, Brower RG, Pronovost PJ. Lung protective mechanical ventilation and two year survival in patients with acute lung injury: prospective cohort study. BMJ. 2012 Apr 5;344:e2124. doi: 10.1136/bmj.e2124. PMID 22491953
- [Background] Needham DM, Dennison CR, Dowdy DW, Mendez-Tellez PA, Ciesla N, Desai SV, Sevransky J, Shanholtz C, Scharfstein D, Herridge MS, Pronovost PJ. Study protocol: The Improving Care of Acute Lung Injury Patients (ICAP) study. Crit Care. 2006 Feb;10(1):R9. doi: 10.1186/cc3948. PMID 16420652
- [Background] Kamdar BB, Huang M, Dinglas VD, Colantuoni E, von Wachter TM, Hopkins RO, Needham DM; National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome Network. Joblessness and Lost Earnings after Acute Respiratory Distress Syndrome in a 1-Year National Multicenter Study. Am J Respir Crit Care Med. 2017 Oct 15;196(8):1012-1020. doi: 10.1164/rccm.201611-2327OC. PMID 28448162
- [Background] Self WH, Grijalva CG, Zhu Y, Talbot HK, Jules A, Widmer KE, Edwards KM, Williams JV, Shay DK, Griffin MR. Emergency department visits for influenza A(H1N1)pdm09, Davidson County, Tennessee, USA. Emerg Infect Dis. 2012 May;18(5):863-5. doi: 10.3201/eid1805.111233. PMID 22516043
- [Background] Tchetgen Tchetgen EJ. Identification and estimation of survivor average causal effects. Stat Med. 2014 Sep 20;33(21):3601-28. doi: 10.1002/sim.6181. Epub 2014 May 29. PMID 24889022
- [Background] Schoenfeld DA, Bernard GR; ARDS Network. Statistical evaluation of ventilator-free days as an efficacy measure in clinical trials of treatments for acute respiratory distress syndrome. Crit Care Med. 2002 Aug;30(8):1772-7. doi: 10.1097/00003246-200208000-00016. PMID 12163791
- [Background] Ramirez JA, Wiemken TL, Peyrani P, Arnold FW, Kelley R, Mattingly WA, Nakamatsu R, Pena S, Guinn BE, Furmanek SP, Persaud AK, Raghuram A, Fernandez F, Beavin L, Bosson R, Fernandez-Botran R, Cavallazzi R, Bordon J, Valdivieso C, Schulte J, Carrico RM; University of Louisville Pneumonia Study Group. Adults Hospitalized With Pneumonia in the United States: Incidence, Epidemiology, and Mortality. Clin Infect Dis. 2017 Nov 13;65(11):1806-1812. doi: 10.1093/cid/cix647. PMID 29020164